CLINICAL TRIAL: NCT02093520
Title: MILD® Percutaneous Image-Guided Lumbar Decompression Versus Epidural Steroid Injections in Patients With Lumbar Spinal Stenosis Exhibiting Neurogenic Claudication
Brief Title: The MiDAS ENCORE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MiDAS ENCORE
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-05

CONDITIONS: Spinal Stenosis, Lumbar Region, With Neurogenic Claudication
Keywords: Lumbar Spinal Stenosis; Spinal Stenosis; Neurogenic Claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MILD (Active Comparator): The MILD procedure is an image-guided minimally-invasive lumbar decompression
  Interventions: Procedure: MILD Procedure
- Epidural Steroid Injection (ESI) (Active Comparator): An epidural steroid injection (ESI) is a combination of a corticosteroid with a local anesthetic pain relief medicine.
  Interventions: Drug: Epidural Steroid Injection

INTERVENTIONS:
Procedure: MILD Procedure — The percutaneous procedure is performed under fluoroscopic guidance to effect a lumbar decompression with minimal surrounding tissue and bone disruption. The mild® Device Kit is utilized to access, capture and remove bone and tissue.
  Other Names: MILD lumbar decompression
  Arms: MILD
Drug: Epidural Steroid Injection — Injection of epidural steroids into the lumbar spine
  Other Names: ESI
  Arms: Epidural Steroid Injection (ESI)

SUMMARY:
Study Objective: To compare patient outcomes following treatment with either the MILD procedure or epidural steroid injections (ESIs) in patients with painful lumbar spinal stenosis exhibiting neurogenic claudication and having verified ligamentum flavum hypertrophy as a contributing factor.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years or older and a Medicare beneficiary.
2. Patients experiencing neurogenic claudication symptoms for at least 3 months duration which has failed to respond or poorly responded to physical therapy, home exercise programs, and oral analgesics.
3. LSS with neurogenic claudication diagnosed via:

   1. Symptomatic diagnosis and
   2. Radiologic evidence of LSS with unilateral or bilateral ligamentum flavum >2.5mm confirmed by pre-op MRI or CT performed within 12 months of baseline visit.
4. Patients with comorbid conditions commonly associated with spinal stenosis, such as osteophytes, facet hypertrophy, minor spondylolisthesis, foraminal stenosis, and/or disk protrusion may be included unless the treating physician has determined that the condition is too advanced.
5. Available to complete 6 month and one year follow-up visits.

Exclusion Criteria:

1. ODI Score < 31 (0-100 ODI Scale).
2. NPRS Score < 5 (0-10 NPRS Scale).
3. Prior surgery at any treatment level.
4. History of recent spinal fractures with current related pain symptoms.
5. Patients with Grade III or higher spondylolisthesis.
6. Motor deficit or disabling back and/or leg pain from causes other than LSS neurogenic claudication (e.g., acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.).
7. Unable to walk ≥ 10 feet unaided before being limited by pain. In this context, 'unaided' means without the use of a cane, walker, railing, wall, another person or any other means of walking assistance.
8. Patients previously randomized and/or treated in this clinical study.
9. Patients that have previously received the MILD procedure.
10. ESI during eight weeks prior to study enrollment.
11. Epidural lipomatosis (if it is deemed to be a significant contributor of canal narrowing by the physician).
12. On (or pending) Workman's Compensation or known to be considering litigation associated with back pain.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramsin Benyamin, MD, Principal Investigator — AAPM; ASIPP; ISIS; ASA; Peter Staats, MD, Principal Investigator — AAPM; ASIPP; ASA
Locations (12):
- United States (12):
  - Synovation Medical Group, Chula Vista, California
  - Spine Intervention Medical Group/Fresno Surgical Hospital, Fresno, California
  - The Spine Institute, Murrieta, California
  - Newport Beach Headache and Pain, Newport Beach, California
  - Millennium Pain Center, Bloomington, Illinois
  - Frankfort Pain Clinic, Frankfort, Kentucky
  - MI Interventional Pain Center, Cherry Island, Michigan
  - Michigan Pain Specialist, Ypsilanti, Michigan
  - Mayo Clinic Pain Management, Rochester, Minnesota
  - Premier Pain, Shrewsbury, New Jersey
  - Southern Spine Institute, Mt. Pleasant, South Carolina
  - SC Spine and Pain Specialists, Myrtle Beach, South Carolina

REFERENCES:
- [Derived] Staats PS, Chafin TB, Golovac S, Kim CK, Li S, Richardson WB, Vallejo R, Wahezi SE, Washabaugh EP 3rd, Benyamin RM; MiDAS ENCORE Investigators. Long-Term Safety and Efficacy of Minimally Invasive Lumbar Decompression Procedure for the Treatment of Lumbar Spinal Stenosis With Neurogenic Claudication: 2-Year Results of MiDAS ENCORE. Reg Anesth Pain Med. 2018 Oct;43(7):789-794. doi: 10.1097/AAP.0000000000000868. PMID 30199512
- [Derived] Benyamin RM, Staats PS, MiDAS Encore I. MILD(R) Is an Effective Treatment for Lumbar Spinal Stenosis with Neurogenic Claudication: MiDAS ENCORE Randomized Controlled Trial. Pain Physician. 2016 May;19(4):229-42. PMID 27228511
- [Derived] Staats PS, Benyamin RM; MiDAS ENCORE Investigators. MiDAS ENCORE: Randomized Controlled Clinical Trial Report of 6-Month Results. Pain Physician. 2016 Feb;19(2):25-38. PMID 26815247

RESULTS

PARTICIPANT FLOW:
Groups:
- Minimally Invasive Lumbar Decompression (MILD): Image guided minimally-invasive lumbar decompression
  Minimally Invasive Lumbar Decompression: The percutaneous procedure is performed under fluoroscopic guidance to effect a lumbar decompression with minimal surrounding tissue and bone disruption. The mild® Device Kit is utilized to access, capture and remove bone and tissue.
Period: Overall Study
Arm/Group | Minimally Invasive Lumbar Decompression (MILD) | Epidural Steroid Injection (ESI)
Started | 149 | 153
Completed | 143 | 131
Not Completed | 6 | 22
Not completed — Not treated | 6 | 22

BASELINE CHARACTERISTICS:
Groups:
- MILD: Image guided minimally-invasive lumbar decompression
  Minimally Invasive Lumbar Decompression: The percutaneous procedure is performed under fluoroscopic guidance to effect a lumbar decompression with minimal surrounding tissue and bone disruption. The mild® Device Kit is utilized to access, capture and remove bone and tissue.
- Total: Total of all reporting groups
Arm/Group | MILD | Epidural Steroid Injection (ESI) | Total
Number analyzed (Participants) | 149 | 153 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.6 (7.0) | 75.0 (7.0) | 75.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 95 | 170
  Male | 74 | 58 | 132
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149 | 153 | 302
ODI [Mean (Standard Deviation); unit: units on a scale] — The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire.
  0 to 20: Minimal disability 21-40: Moderate Disability 41-60: Severe Disability 61-80: Crippling back pain 81-100: These patients are either bed-bound or have an exaggeration of their symptoms.
  units on a scale | 53.0 (12.9) | 51.7 (12.0) | 52.3 (12.4)
NPRS [Mean (Standard Deviation); unit: units on a scale] — The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  units on a scale | 7.7 (1.4) | 7.8 (1.3) | 7.8 (1.4)
ZCQ [Mean (Standard Deviation); unit: units on a scale] — The Zurich Claudication Questionnaire (ZCQ) is a disease-specific self-report outcome. The ZCQ quantifies severity of symptoms, physical function characteristics, and patient's satisfaction after treatment. The scale relates to symptoms over the past month.
  ZCQ consists of three subscales:
  1. Symptom severity scale (questions I-VII) Possible range of the score is 1 to 5.
  2. Physical function scale (questions VIII-XII): Possible range of scores is 1 to 4.
  3. Patient's satisfaction with treatment scale (questions XIII-XVIII): the range of the scale is 1 to 4.
  units on a scale
    Symptom Severity | 3.5 (0.5) | 3.5 (0.6) | 3.5 (0.6)
    Physical Function | 2.9 (0.5) | 2.8 (0.4) | 2.8 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Clinically Significant Improvement in the Oswestry Disability Index at 12 Months
Description: Proportion of ODI Responders from baseline to one year follow-up in the treatment group versus the proportion of ODI Responders from baseline to one year follow-up in the control group. ODI Responders are defined as those patients achieving the validated Minimal Important Change in ODI score from baseline to follow-up as a clinically significant efficacy threshold.
Time Frame: 12 months
Population: Six participants in the MILD and 22 in the ESI group did not receive study treatment, therefore 143/149 MILD participants and 129/153 ESI participants were analyzed for outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Lumbar Decompression (MILD) | Epidural Steroid Injection (ESI)
Number analyzed (Participants) | 143 | 129
Participants | 83 | 35

2. Secondary Outcome: Number of Participants Who Acheived a Clinical Significant Improvement in the Numeric Pain Rating Scale (NPRS) at 12 Months
Description: Proportion of NPRS Responders from baseline to one year follow-up in each of the two treatment groups using validated Minimal Important Change value as the clinically significant efficacy threshold.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Lumbar Decompression (MILD) | Epidural Steroid Injection (ESI)
Number analyzed (Participants) | 143 | 129
Participants | 82 | 35

3. Secondary Outcome: Number of Participants Who Achieved a Clinically Significant Improvement in the Zurich Claudication Questionnaire (ZCQ) at 12 Months
Description: Proportion of ZCQ Responders from baseline to one year follow-up in each of the two treatment groups using validated Minimal Important Change value as the clinically significant efficacy threshold.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Minimally Invasive Lumbar Decompression (MILD) | Epidural Steroid Injection (ESI)
Number analyzed (Participants) | 143 | 129
Participants
  Symptom Severity | 74 | 41
  Physical Function | 63 | 23
  Patient Satisfaction | 88 | 43

ADVERSE EVENTS:
Description: For standardization of reporting, all adverse events have been coded by an outside agency into MedDRA System Organ Class and Preferred Term classifications
Arm/Group | Minimally Invasive Lumbar Decompression (MILD) | Epidural Steroid Injection (ESI)
All-Cause Mortality (participants affected / at risk) | 2/149 | 0/153
Serious Adverse Events (participants affected / at risk) | 18/149 | 13/153
Other Adverse Events (participants affected / at risk) | 2/149 | 2/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimally Invasive Lumbar Decompression (MILD) (N=149) | Epidural Steroid Injection (ESI) (N=153)
Cardiac Disorders (Cardiac disorders) | 6 (6) | 5 (5)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions (General disorders) | 0 (0) | 2 (2)
Infections and infestations (Infections and infestations) | 5 (5) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) | 4 (6)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecifie (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimally Invasive Lumbar Decompression (MILD) (N=149) | Epidural Steroid Injection (ESI) (N=153)
Cardiac disorders (Cardiac disorders) | 0 (0) | 1 (1) — Procedure related adverse event
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Procedure related adverse event
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) — Procedure related adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No